## **Informed Consent**

Comparative study of two hemodialysis catheter exit site dressing regimens: chlorhexidine gluconate dressing vs chlorhexidine 2% solution.

**Identifier:** NCT05855616 Unique Protocol ID: HUMV-PIE2020-02

Date: 20 september 2021

## **Informed Consent**

Date and signature:

- **Project Title**: Comparative study of two hemodialysis catheter exit site dressing regimens: chlorhexidine gluconate dressing vs chlorhexidine 2% solution.
- **Referral center**: Nephrology Department Hospital Universitario Marqués de Valdecilla

| Ι ( | Name and Surname | ) |
|-----|------------------|---|
|-----|------------------|---|

- I have read the information document accompanying this consent (Information Sheet).
- I have been able to ask questions about the study
- I have received sufficient information about the study
- I have spoken with......
- I understand that my participation is voluntary and I am free to participate or not in the study
- I understand that I can withdraw from the study:
  - Whenever you want
  - Without having to explain myself
  - o Without any impact on the care of my family member.
- I have been informed that all data obtained in this study will be confidential
  and will be treated in accordance with the Regulation (EU) 2016/679 of the
  European Parliament and of the Council of 27 April 2016 on Data Protection
  (GDPR) and the organic law 3/2018 of December 5, on the protection of
  personal data and guarantee of digital rights.

Therefore, I freely give my consent to participate in the study and consent to the access and use of my data under the conditions detailed in the information sheet.

| | Participant's signature | Professional's signature |
|---|---|---|
| | , , | J |
| | Name and surname: | Name and surname: |
| | Date: | Date: |
| In case of revo | cation of Consent: | |
| I, Mr./Ms | | I withdraw |
| the consent given for my participation in the above mentioned study | | |